CLINICAL TRIAL: NCT07015047
Title: Effects of Magnesium L-Threonate on Sleep, Recovery, and Athletic Performance in UCLA Athletes: A Randomized, Placebo-Controlled Trial
Brief Title: Effects of Magnesium L-Threonate on Sleep, Recovery, and Athletic Performance in Collegiate Athletes
Acronym: MgT-Athletes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Jeremy Swisher, MD, Health Sciences Assistant Clinical Professor, Department of Orthopaedic Surgery - Sports Medicine, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB-25-1201
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Recovery of Function (G11.427.698.620); Athletic Performance; Heart Rate Variability (HRV)
Keywords: Magnesium L-Threonate; Sleep Quality; WHOOP; Athlete Recovery; HRV; NCAA Athletes; Sports Medicine; Wearable Technology
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — threonic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnesium L-Threonate (Experimental): Participants assigned to this arm will take 1 gram of magnesium L-threonate (Magtein) in capsule form each evening for 4 weeks. They will wear a WHOOP strap continuously to collect sleep and recovery metrics and complete baseline/follow-up performance testing.
  Interventions: Dietary Supplement: Magnesium L-Threonate
- Placebo (Placebo Comparator): Participants assigned to this arm will take an identical-looking placebo capsule each evening for 4 weeks. They will wear a WHOOP strap continuously to collect sleep and recovery metrics and complete baseline/follow-up performance testing.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Magnesium L-Threonate — Participants in this arm will take 1 gram of magnesium L-threonate (Magtein), provided in capsule form, once daily in the evening for 4 weeks. This supplement is known for its ability to cross the blood-brain barrier and may enhance sleep architecture, autonomic recovery, and cognitive function.
  Arms: Magnesium L-Threonate
Other: Placebo — Identical-looking inert capsule taken nightly for 4 weeks. Used as a comparator to magnesium L-threonate to assess changes in sleep, recovery, and performance metrics.
  Arms: Placebo

SUMMARY:
This study is testing whether a special form of magnesium called magnesium L-threonate can help improve sleep quality, recovery, and physical performance in college athletes. Magnesium is important for muscle recovery and sleep, but many forms of it do not enter the brain well. Magnesium L-threonate is unique in that it can cross the blood-brain barrier and may improve deep and REM sleep, heart rate variability, and brain recovery.

In this study, healthy UCLA varsity athletes aged 18 to 35 will be randomly assigned to take either magnesium L-threonate or a placebo each evening for 4 weeks. They will wear a WHOOP strap to track sleep, recovery, and heart rate data. Performance tests including jump height, grip strength, and reaction time will be completed before and after the 4-week period.

This study will help researchers determine if this supplement can support recovery and training in athletes and whether wearable technology can help monitor these changes in real time.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled trial examining the effects of magnesium L-threonate (MgT) supplementation on sleep architecture, autonomic recovery, and physical performance in collegiate athletes. Magnesium is a critical mineral for neuromuscular and autonomic function, but common forms have limited central nervous system penetration. MgT crosses the blood-brain barrier and has been shown in non-athletic populations to improve sleep depth, REM sleep, and cognitive function. No prior studies have evaluated its effects in athletes.

Approximately 100 UCLA varsity athletes aged 18-35 will be randomized in a 1:1 ratio to receive 1 gram of MgT or placebo nightly for 4 weeks. Participants will wear a WHOOP strap to continuously monitor deep sleep, REM sleep, heart rate variability, resting heart rate, and recovery score. Daily surveys will track subjective sleep quality, recovery, and for female athletes, menstrual phase and symptoms. Performance outcomes including countermovement jump height, handgrip strength, and light-based reaction time will be measured before and after the intervention.

Primary outcomes include objective changes in sleep stages and HRV. Secondary outcomes include changes in physical performance and subjective recovery. This study will provide insight into whether brain-targeted magnesium supplementation can enhance recovery and performance in an athletic population.

ELIGIBILITY:
Inclusion Criteria:

* • Age 18-35 years

  * Current UCLA varsity athlete (any sport)
  * Actively training or competing during the study period
  * Willing to wear a WHOOP strap continuously for 4 weeks
  * Willing to ingest a nightly capsule for 4 weeks
  * Able to provide informed consent and comply with study procedures

Exclusion Criteria:

* • Current use of magnesium supplements or investigational drugs

  * Use of prescription or over-the-counter sleep medications
  * Diagnosed sleep disorder (e.g., insomnia, sleep apnea)
  * Major medical condition limiting training or participation
  * Pregnancy or breastfeeding
  * Known history of chronic kidney or liver disease
  * Allergy or intolerance to magnesium
  * Inability to comply with study procedures (e.g., wearing WHOOP or completing surveys)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Change in Deep Sleep Duration (minutes) from Baseline to Week 4 | Baseline to Week 4
  Deep (slow-wave) sleep duration will be measured nightly using WHOOP wearable sensors. Average weekly deep sleep duration will be calculated and compared between groups.
Change in Heart Rate Variability (HRV) from Baseline to Week 4 | Baseline to Week 4
  HRV (measured in ms) will be captured nightly via WHOOP device. Weekly averages will be analyzed to assess autonomic recovery across time points.

SECONDARY OUTCOMES:
Change in Countermovement Jump Height (cm) from Baseline to Week 4 | Baseline and Week 4
  Jump height will be assessed using force plate technology.
Change in Reaction Time (ms) from Baseline to Week 4 | Baseline and Week 4
  Reaction time will be measured using a standardized light-based reaction test (e.g., BlazePod). Group differences will be analyzed after 4 weeks of supplementation.
Change in Handgrip Strength from Baseline to Week 4 | Baseline and Week 4
  Grip strength will be measured using a calibrated handheld dynamometer. The average value from three trials on the dominant hand will be recorded and analyzed.
Change in Subjective Sleep Quality Score from Baseline to Week 4 | Daily for 4 Weeks (averaged weekly)
  Participants will complete a Single-Item Sleep Quality Scale (rated 0-10) each morning via REDCap. Weekly averages will be used to assess within- and between-group changes.

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA, Los Angeles, California, United States